CLINICAL TRIAL: NCT05675527
Title: Outcomes Following Single Injections of Low-dose Platelet-rich Plasma (PRP), High-dose PRP, or Saline in Patients With Glenohumeral OA: a Randomized Controlled Trial
Brief Title: PRP for Glenohumeral Osteoarthritis
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2022-0720
Record Dates: First submitted 2022-12-28; First posted 2023-01-09 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Shoulder Osteoarthritis
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Low-dose PRP (Experimental): Patients will receive a single injection of 6 ml low-dose platelet-rich plasma (PRP) into the glenohumeral joint. Low-dose is defined as a platelet yield of 3X (i.e., 3-fold increase in platelets in PRP compared to whole blood).
  Interventions: Biological: Low-dose PRP
- High-dose PRP (Experimental): Patients will receive a single injection of 6 ml high-dose platelet-rich plasma (PRP) into the glenohumeral joint. High-dose is defined as a platelet yield of 12X (i.e., 12-fold increase in platelets in PRP compared to whole blood).
  Interventions: Biological: High-dose PRP
- Saline control (Placebo Comparator): Patients will receive a single injection of 6 ml saline into the glenohumeral joint.
  Interventions: Other: Saline

INTERVENTIONS:
Biological: Low-dose PRP — Injection
  Arms: Low-dose PRP
Biological: High-dose PRP — Injection
  Arms: High-dose PRP
Other: Saline — Injection
  Arms: Saline control

SUMMARY:
The glenohumeral joint is the third most common large joint to be affected by OA. Conservative treatments include physical activity, corticosteroid injections, and medications. PRP is an emerging treatment that has shown efficacy in different musculoskeletal conditions. The use of PRP for glenohumeral OA has been described sparingly in the literature but has shown efficacy in a couple studies and case reports. However, all of the previous studies investigating PRP for glenohumeral OA have focused on low-dose PRP preparations (~3X), and none have compared PRP treatment to saline treatment. This study aims to compare outcomes following single injections of low-dose PRP, high-dose PRP, or saline in patients with glenohumeral osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* 18-100 years old
* Average NRS pain greater than or equal to 5/10 as a direct result of glenohumeral osteoarthritis (any severity: mild, moderate, or severe) and/or chondral lesion or loss
* At least 3 months of pain after onset of symptoms that has failed conservative treatments, including physical therapy
* MRI of the affected joint
* Transient relief of symptoms after a diagnostic intra-articular injection into the joint
* Email address or network access

Exclusion Criteria:

* Inability to hold non-steroidal anti-inflammatory drugs for 2 weeks prior and 1 month after the injection
* Prior platelet-rich plasma injection
* Steroid injection within 3 months of the initial injection
* Hyaluronic acid within 6 months of the initial injection
* Involved in workers' compensation or active litigation involving the affected joint
* History of Plavix use
* Known uncontrolled systemic illness (uncontrolled diabetes, HIV, vasculitis, autoimmune/autoinflammatory disease)
* Presence of acute fractures or gross mechanical deformities
* Concurrent "uncontrolled" cervical disorders

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2023-05-02 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
American Shoulder and Elbow Surgeons (ASES) Shoulder Score | 3 months post-injection
  The ASES measures pain and function in activities of daily living related to the shoulder. On a 100-point scale, a higher score represents less pain/higher function.

SECONDARY OUTCOMES:
Average numerical rating scale (NRS) pain score | Up to 12 months post-injection
  Average NRS pain during the past week. This is on a scale of 0-10, with 0 representing no pain and 10 representing the worst pain possible.
Patient-Reported Outcomes Measurement Information System (PROMIS)-10 Global Health measure | Up to 12 months post-injection
  The PROMIS-10 assesses physical health and mental health. A higher score represents better physical health and mental health.
PROMIS-Upper Extremity computer adaptive test (CAT) | Up to 12 months post-injection
  The PROMIS-Upper Extremity CAT measures upper extremity (shoulder) function. A higher scores represents better function.
Medication use | Up to 12 months post-injection
  Patients will be asked if they are using any of the following medications: non-steroidal anti-inflammatory drugs, opioids, selective serotonin reuptake inhibitors, or neuropathic medications.
PROMIS Sleep Disturbance | Up to 12 months post-injection
  The PROMIS sleep disturbance measures sleep impairment/disturbance. A higher score represents more sleep disturbance (e.g., worse sleep quality).
Patient satisfaction | Up to 12 months post-injection
  Patient satisfaction is assessed on a 0-10 scale, with 0 meaning "not satisfied at all" and 10 meaning "very satisfied".

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital for Special Surgery, New York, New York, United States